CLINICAL TRIAL: NCT00262509
Title: Emergency Egress and Information System for Persons With Vision Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention worsened performance for first 17 of 24 planned participants.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: C3905-R
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Blindness
Keywords: Rehabilitation; Sensory Aid
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egress Badge Performance (Experimental): Blind subjects are walked into a building to a specific location, and then are asked to find their way out of the building.
  Interventions: Device: Egress Badge
- Baseline Egress Performance (No Intervention): Blind subjects are walked into a building to a particular location and then asked to find their way out of the building.

INTERVENTIONS:
Device: Egress Badge — Egress Badge is worn by subjects who are asked to use the badge to exit the building. The badge indicates the direction of each exit sign on route to an exit.
  Arms: Egress Badge Performance

SUMMARY:
The purpose of the research project is to develop and evaluate an emergency egress system for persons with visual impairment, which would use existing lighted exit signage to provide egress information at a distance of up to 100 feet.

DETAILED DESCRIPTION:
The purpose of the proposed three-year research project is to develop and evaluate an emergency egress system for persons with visual impairment. This system would use existing lighted exit signage to provide egress information at a distance of up to 100 feet. The distance is the same as the required visibility distance of lighted exit signs for sighted persons. By offering egress information at an equivalent distance, the investigators hypothesize that people with visual impairment can approach the egress performance of sighted persons.

The information transmitted will be equivalent to what a sighted person obtains, namely, the direction of the exit door. In addition, a description of the exit route will be provided including the distance to the exit door; lighting conditions, hazards and obstacles that will be encountered on the exit route; the distance down to the street; and where on the street they will be when they get out of the building. A receiver worn by the person will include a tiny optical array to sense the direction of each exit sign. The receiver will also translate the transmitted signal into a spoken message. A low-profile stereo bone conduction headset will indicate the direction to each exit sign along a path to the exit door. For people with some hearing loss, this same low-profile headset will be used to simulate a light "tap" to one side or other of the head to indicate direction. Such directional "tapping" output may also prove effective when loud alarms are blaring.

The objectives are to:

1. develop Talking Exit Lights with a range of at least 100 feet,
2. write software for the user device to accurately indicate the direction of Talking Exit Lights and provide spoken messages,
3. optimize the user interface to make it easy and intuitive to use,
4. test the accuracy and reliability of the developed system in terms of transmission range and directional accuracy, and
5. conduct subject evaluations of the new system.

Two versions of transmitting exit signs will be developed:

1. a retro-fit design for existing fluorescent light exit signs, and
2. a Light Emitting Diode (LED) design for the LED exit signs now going into newly constructed buildings.

For the retro-fit version, Talking Lights, LLC, will modify the physical shape and size of their Talking Light digital ballast, making it a fully compatible replacement for existing exit sign ballasts. VA investigators will develop the LED version, designing and constructing a microprocessor-controlled system for storing and transmitting information using LEDs. Both designs will use secure power line communications to upload transmittal information to specific exit signs, each of which will have its own ID number. Finally, VA investigators will write software for the existing Talking Lights PocketPC receiver to interpret sensor signals, obtain sign location data, and convert this data into a stereo sound presentation of exit sign direction.

This development will be accomplished via a Cooperative Research and Development Agreement (CRADA) with Talking Lights LLC, which holds a patent on an electronic ballast that converts standard fluorescent bulbs into digital information transmitters. The company will also provide a PocketPC receiver that decodes their proprietary transmission signal, and a 5-sensor optical array capable of picking up their signal over a 150-degree field. As part of this CRADA, Talking Lights will modify their ballast to match the form-factor of ballasts in exit signs. Further, they will release their proprietary encoder design to VA investigators so that the LED Exit Light design can be made fully compatible with the fluorescent light design.

Once developed and optimized, investigators hypothesize a dramatic improvement in egress performance for all ages of two populations:

1. people with severe vision loss who use a white cane or dog for mobility, and
2. people with low vision who do not use a white cane or dog for mobility, yet have problems reading and locating exit signs.

Results will be published and presented for review to the National Fire Prevention Agency (NFPA) for consideration as part of the Life Safety Code, and to the Building Officials and Code Administrators (BOCA) for consideration as part of the National Building Code.

COMPARISONS: Egress using existing emergency exit signage.

ELIGIBILITY:
Inclusion Criteria:

* Must Be Blind with no better vision than light perception
* Must be able to walk the necessary distances, i.e., three hours of intermittent indoor walking
* OMCT (Orientation-Memory Concentration Test) of 10 or less

Exclusion Criteria:

* Patients currently being treated at Atlanta VA Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Ross, MSEE Med, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from July through September, 2009. They were recruited from the VA Medical Center Eye Clinic and the Atlanta Center for Visual Impairment.
Pre-assignment Details: 17 participants recruited after 23 potential participants contacted by phone from our VA subject registry. Of the 23 contacted, 3 screened out as not meeting inclusion criteria, and 3 chose not to participate.
Groups:
- Baseline First, Then Intervention: Baseline First: For two separate timed trials Blind Participants are walked into a building to different randomized locations, and then asked to find their way out of the building. Each Trial lasted at most 15 minutes.
  Intervention Next: Blind Participants are trained for 15 minutes in the use of the egress badge, then in two separate timed trials are walked into a building to different randomized locations, and are asked to find their way out of the building. Each Trial lasted at most 15 minutes.
- Intervention First, Then Baseline: Intervention First: Blind Participants are trained for 15 minutes in the use of the egress badge, then in two separate timed trials are walked into a building to different randomized locations, and are asked to find their way out of the building. Each Trial lasted at most 15 minutes.
  Baseline Next: For two separate timed trials Blind Participants are walked into a building to different randomized locations, and then asked to find their way out of the building. Each Trial lasted at most 15 minutes.
Period: Overall Study
Arm/Group | Baseline First, Then Intervention | Intervention First, Then Baseline
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes groups randomized to do either baseline tests first or Intervention tests first
Groups:
- First Baseline, Then Intervention: Baseline First: For two separate timed trials Blind Participants are walked into a building to different randomized locations, and then asked to find their way out of the building. Each Trial takes at most 15 minutes.
  Intervention Next: Blind Participants are trained for 15 minutes in the use of the egress badge, then in two separate timed trials are walked into a building to different randomized locations, and are asked to find their way out of the building. Each Trial takes at most 15 minutes.
- First Intervention, Then Baseline: Intervention First: Blind Participants are trained for 15 minutes in the use of the egress badge, then in two separate timed trials are walked into a building to different randomized locations, and are asked to find their way out of the building. Each Trial takes at most 15 minutes.
  Baseline Next: For two separate timed trials Blind Participants are walked into a building to different randomized locations, and then asked to find their way out of the building. Each Trial takes at most 15 minutes.
- Total: Total of all reporting groups
Arm/Group | First Baseline, Then Intervention | First Intervention, Then Baseline | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.78 (10.72) | 52.75 (7.07) | 50.12 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Time to Exit Building
Description: Subjects are walked into a building to a specific location and then asked to find their way out of the building. Time to Exit Building is measured. This is protocol is performed twice, and the times averaged to obtain the outcome measure.
Time Frame: 30 minutes total, 15 minutes for each of two timed trials
Population: Total number of participants completing study
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Egress Time
Groups:
- Intervention: All Blind Participants are trained for 15 minutes in the use of the egress device, then for two separate trials are walked into a building to a specific location, and are asked to find their way out of the building. Their egress performance is timed for each trial. The outcome measure is obtained by averaging the two trial times
- Baseline: All Blind Participants, in two separate trials, are walked into a building to a specific location, and then are asked to find their way out of the building. Their egress performance is timed for each trial. The outcome measure is calculated as the average of the trial times.
Arm/Group | Intervention | Baseline
Number analyzed (Participants) | 17 | 17
Number analyzed (Egress Time) | 17 | 17
seconds | 198 (47) | 165 (63)

ADVERSE EVENTS:
Time Frame: 2.5 hours per subject during the intervention and baseline trials
Groups:
- Egress Badge Intervention: Blind Participants are trained for 15 minutes in the use of the egress badge, then for two separate trials they are walked into a building to a different locations, and are asked to find their way out of the building.
- Baseline Egress: Blind subjects are walked into a building to different locations in two separate trials and then asked to find their way out of the building.
Arm/Group | Egress Badge Intervention | Baseline Egress
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
Trials were terminated early with just 17 Participants of the planned 24, as the intervention was NOT providing measurable benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No